CLINICAL TRIAL: NCT03854734
Title: A Randomized Study to Determine the Efficacy of a Multi-tiered Community- and School-based Approach to Enhance School-aged Children's Recommended Vaccinations.
Brief Title: Healthy, Immunized Communities Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jennifer Kraschnewski, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Study000011289
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Vaccine Hesitancy; Communicable Diseases in Children
Keywords: Vaccinations; Vaccine hesitancy; School-based research
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Following collection of baseline data, schools will be randomized. Study staff measuring the primary outcome will be blinded to school group assignment. Given the intervention, it is not possible to blind participants to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Educational emails about broad health topics to keep control group engaged
- Multi-Component Intervention (Active Comparator): (1) a community event to raise parental awareness of the importance of vaccination; (2) social marketing to target parents' attitudes and knowledge around vaccinations in the form of educational material
  Interventions: Behavioral: Community Event; Behavioral: Educational Material

INTERVENTIONS:
Behavioral: Community Event — Formative focus group data was used to design an educational community event to improve information share and vaccine education/knowledge.
  Arms: Multi-Component Intervention
Behavioral: Educational Material — Formative focus group data was used to design educational messaging to be electronically distributed to intervention participants
  Arms: Multi-Component Intervention

SUMMARY:
This project aims to understand how improving vaccine education and awareness can impact the number of parents who vaccinate, or intend to vaccine, their middle school-aged children with age-appropriate vaccines, including human papillomavirus (HPV), meningitis (MCV) and tetanus, diphtheria, pertussis (TDap).

DETAILED DESCRIPTION:
Vaccines are considered one of the greatest public health successes. Unfortunately, an increasing rate of parental resistance in recent years has led to a reemergence of vaccine-preventable diseases. This project seeks to determine the effect of a multi-tiered school and community-based approach to improving rates of parental intent to vaccinate for middle school-aged vaccinations including Human Papillomavirus (HPV), meningitis (MCV) and Tetanus, Diphtheria, Pertussis (TDap).

By randomizing participating schools, parents receiving the intervention participated in (1) a community-based event to raise parental awareness of the importance of vaccination and (2) a social marketing campaign targeting parents' attitudes and knowledge around vaccinations.

The Investigators hypothesized that participation in this study would increase parental intention to vaccinate. In addition, this study intended to improve rates of recommended vaccination among middle school-aged children, as measured through vaccine uptake information required for annual entry into Pennsylvania public schools.

The Penn State team brings a breadth of experience in pediatrics, community-engaged research, adolescent health, and engagement with schools.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Parents and guardians of children who attend a School District of Lancaster middle schools
* Individuals who read and understand English
* Individuals with an email address

Exclusion Criteria

* Individuals who are non-English speaking
* Parents/Guardians <18 years or older who do not have children attending a middle school in the School District of Lancaster
* Individuals who do not have an email address
* Individuals who plan on moving out of the Lancaster City area in the next year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kraschnewski, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The following steps will be taken to protect subjects' privacy interests: identification and recruitment of potential subjects follows procedures consistent with privacy standards; consent discussion and research interventions will take place in a private setting; the information being collected will be limited to only the minimum amount of data necessary to accomplish the research purposes; the people with access to the identifiable research data will be limited to the minimum necessary as specified in the application and consent process. To external researchers or sponsors, data will be sent sent/received in aggregate/metrics (just counts, no individual data).

REFERENCES:
- See also: Peer-reviewed manuscript describing primary study outcomes — https://doi.org/10.1016/j.jvacx.2023.100273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between February and September 2019. Participants were recruited through the participating school partner, who distributed a recruitment flyer via email and through social media channels. Participants were also recruited through in-person events at the participating schools, such as chorus concerts and parent-teacher conferences.
Pre-assignment Details: Four schools were randomized to two arms (intervention vs. control). 502 individuals were assessed for eligibility and 354 were excluded for not meeting inclusion criteria (n=265) or declining to participate (n=89).
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | Usual Care | Multi-Component Intervention
Started | 70; 2 Schools | 78; 2 Schools
Completed | 70; 2 Schools | 78; 2 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Multi-Component Intervention | Total
Number analyzed (Participants) | 70 | 78 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.00 (9.79) | 40.46 (8.59) | 39.32 (9.21)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 11 | 7 | 18
  Gender: Female | 57 | 68 | 125
  Gender: No response | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 32 | 43 | 75
  Race/Ethnicity: Black/African American | 6 | 7 | 13
  Race/Ethnicity: Hispanic or Latino | 22 | 20 | 42
  Race/Ethnicity: Other | 10 | 7 | 17
  Race/Ethnicity: No response | 0 | 1 | 1
Relationship Status [Count of Participants; unit: Participants]
  Single OR separated OR divorced OR widowed | 26 | 30 | 56
  Married OR living with partner | 43 | 46 | 89
  No response | 1 | 2 | 3
Annual household income [Count of Participants; unit: Participants]
  ≤$40,000 | 31 | 27 | 58
  $40,001 - $80,000 | 26 | 25 | 51
  >$80,000 | 12 | 23 | 35
  No Response | 1 | 3 | 4
Education [Count of Participants; unit: Participants]
  High School or Less | 35 | 29 | 64
  Some College | 15 | 12 | 27
  College Graduate | 20 | 37 | 57
  No response | 0 | 0 | 0
Relationship to child [Count of Participants; unit: Participants]
  Mother | 56 | 66 | 122
  Father | 9 | 8 | 17
  Guardian/Grandparent | 5 | 4 | 9
Grade of child [Count of Participants; unit: Participants]
  6th | 37 | 33 | 70
  7th | 22 | 29 | 51
  8th | 11 | 16 | 27
Gender of child [Count of Participants; unit: Participants]
  Male | 40 | 44 | 84
  Female | 30 | 34 | 64
Parent participation in school events per year [Count of Participants; unit: Participants]
  ≤1 | 41 | 37 | 78
  2-5 | 25 | 24 | 49
  ≥6 | 4 | 16 | 20
  No response | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Intent to Vaccinate Adolescent Child (Tdap, MCV, HPV)
Description: Parental intent to vaccinate their adolescent child with Tdap, MCV, and HPV vaccines, was dichotomized for each vaccine in the survey. Tdap and MCV included the options 1) intention to vaccinate/vaccinated ("plan to get this shot before the first day of 7th grade" or "up-to-date with this shot") or 2) no intention to vaccinate ("no plans to get this shot" or "have or plan to submit an exemption for this shot"). The HPV variable excluded the option "have or plan to submit an exemption for this shot" as vaccine is not required for school entry. Variables (Tdap, MCV, HPV) were compared within and between treatment groups from baseline to 6 mo. follow up with a generalized estimating equations model using the framework of a log-binomial logistic regression model. Risk ratios resulting from these models were used to quantify the magnitude and direction of any significant differences.
Time Frame: Participants were assessed at baseline and follow-up at 6 months.
Population: 4 middle schools were randomized to either a usual care or multi-component intervention arm. Participants (parents) were assigned to a study arm based on their associated middle school. 30 participants either did not complete the follow up survey (n=27) or did not answer all questions (n=3), as questions were not required. Discrepancies in percentage reporting in the outcomes table below results from inconsistent rates of missingess (range 0-4) across variables (Tdap, MCV, HPV).
Measure: Number; unit: percentage of participants
Units Other Than Participants: Middle Schools
Arm/Group | Usual Care | Multi-Component Intervention
Number analyzed (Participants) | 70 | 78
Number analyzed (Middle Schools) | 2 | 2
percentage of participants
  Tetanus, diphtheria, acellular pertussis (Tdap) : Vaccine intention at baseline | 74.3 | 83.3
  Tetanus, diphtheria, acellular pertussis (Tdap) : Vaccine intention at follow-up | 97.9 | 93.0
  Meningococcal conjugate vaccine (MCV) : Vaccine intention at baseline | 72.9 | 80.5
  Meningococcal conjugate vaccine (MCV) : Vaccine intention at follow-up | 91.5 | 91.6
  Human papillomavirus (HPV) : Vaccine intention at baseline | 84.1 | 84.4
  Human papillomavirus (HPV) : Vaccine intention at follow-up | 85.7 | 87.3
Statistical Analysis 1: Comparison: Multi-Component Intervention; Analysis for vaccine intention of Tdap; Test type: Superiority — Generalized estimating equations (GEE) model using the framework of a log-binomial logistic regression model; Regression, Logistic; Risk Ratio (RR) = 1.12, 95% CI 2-sided [1.00 to 1.25]
Statistical Analysis 2: Comparison: Multi-Component Intervention; Analysis for vaccine intention of MCV; Test type: Superiority — Generalized estimating equations (GEE) model using the framework of a log-binomial logistic regression model; Regression, Logistic; Risk Ratio (RR) = 1.14, 95% CI 2-sided [1.00 to 1.29]
Statistical Analysis 3: Comparison: Multi-Component Intervention; Analysis for vaccine intention of HPV; Test type: Superiority — Generalized estimating equations (GEE) model using the framework of a log-binomial logistic regression model; Regression, Logistic; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.96 to 1.14]

ADVERSE EVENTS:
Time Frame: Due to the nature of the intervention, adverse events were not monitored/assessed.
Description: Due to the nature of the intervention, adverse events were not monitored/assessed.
Arm/Group | Usual Care | Multi-Component Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We experienced low parent participation in the intervention activities, potentially limiting the effectiveness of the intervention and resulting outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03854734/Prot_SAP_000.pdf